CLINICAL TRIAL: NCT03741374
Title: Analysis of Intrabony Defects Treated With Minimally-invasive Non-surgical Therapy: A Prospective Cohort Multicentre Study
Brief Title: Minimally-invasive Non-surgical Therapy of Intrabony Defects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Ravenscourt Dental Practice (Unknown); South Coast Dental Specialists (Unknown); Claremonth Dental Practice (Unknown); Pall Mall Dental (Other); Rose Lane Dental Practice (Unknown); Periosouth (Unknown); Clinica de Periodoncia (Unknown); Studio Dentistico Associato Montevecchi D' Alessandro (Unknown); 11th floor 141 Queen St. Brisdane (Unknown); The Dentist (Other); High Barnet Dental Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QMERC 2018/56
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally-invasive non-surgical therapy (Experimental): Intrabony defects treated with Minimally-invasive non-surgical therapy (MINST)
  Interventions: Procedure: Minimally-invasive non-surgical therapy (MINST)

INTERVENTIONS:
Procedure: Minimally-invasive non-surgical therapy (MINST) — A non-surgical minimally-invasive treatment protocol, named MINST, has been proposed (Ribeiro et al. 2011) for the treatment of periodontitis, in order to minimise patient discomfort and maximise the healing potential. This technique usually involve the use of magnification lenses or microscopes and small instruments which would reduce the risk of tissue trauma compared with traditional instruments.

SUMMARY:
This investigation aims to assess the clinical and radiographic outcomes of intrabony defects treated with minimally-invasive non-surgical therapy.

DETAILED DESCRIPTION:
Periodontal diseases are inflammatory conditions that affect the supporting apparatus of the teeth, including gingiva and alveolar bone. The bone loss resulting from periodontitis often is irregular and localised, giving onset to 'intrabony' or 'vertical defects' affecting one side of the tooth more than the other and more than on the neighbouring teeth. Periodontal intrabony defects have been associated with a higher risk of further progression and eventually tooth loss.

The treatment of periodontitis involves a non-specific reduction of the bacterial load below the gingival margin. This is achieved by oral hygiene instructions (OHI) and non-surgical periodontal therapy (NSPT), aimed at removing calculus and disrupting the plaque biofilm from the affected root surfaces. Intrabony defects are considered sites requiring therapy, often beyond NSPT. Decades ago, intrabony defects were treated with surgical elimination of the defect achieved by sacrificing the adjacent healthy supportive or non-supportive bone. More recently periodontal regenerative procedures have been advocated for deep intrabony defects, which are considered amenable for guided tissue regeneration. This technique results in regeneration of periodontal attachment measurable histologically and radiographically and measurable clinically. However, this is associated with potential morbidity and high costs due to the use of bone graft and barrier materials and is not always predictable. The more recent introduction of minimally-invasive surgical therapy (MIST), modified-MIST (M-MIST) and single-flap approach suggested that the use of biomaterials may not be so crucial for obtaining periodontal regeneration.

A retrospective study from our group has shown that non-surgical periodontal treatment of intrabony defects results in clinical improvements (measured as PPD reductions and clinical attachment level-CAL- gain) but also in bone fill of the bony defects, measurable radiographically. The extent of the radiographic resolution of the defect was positively associated with initial defect depth and use of adjunctive antibiotics, while smoking seemed to negatively influence this outcome. A non-surgical minimally-invasive treatment protocol, named MINST, has been proposed along these principles. A more recent retrospective analysis has revealed a reduction in bony defect of nearly 3 mm for cases treated with minimally-invasive non-surgical therapy. The effect of MINST may be mediated by improved blood flow and stable blood clot in the intrabony defect. However, very few studies have been published on MINST and no data are available on generalizability and wide applicability of MINST.

This is a prospective cohort multicentre study to assess the effect of a modified minimally-invasive non-surgical therapy (MINST) approach in the healing of 100 periodontal intrabony defects in patients with periodontitis seen in private practice. The therapists responsible for delivering this treatment as part of this study all have experience in routinely carrying out this or similar procedures for this type of periodontal defects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Diagnosis of Periodontitis (Tonetti et al. 2018)
3. Presence of ≥1 'intrabony defect' (PPD and CAL >5 mm with radiographic intrabony defect depth ≥3mm and not in a site associated with furcation involvement)
4. Signed informed consent [Participants must be able and willing to read and sign a copy of the "Informed Consent Form" (ICF) form after reading the "Patient Information Leaflet" (PIS), and after the nature of the study has been fully explained].

Exclusion Criteria:

1. Smoking (current or in past 5 years, including electronic cigarettes, vaping or similar)
2. Medical history including diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases
3. Presence of drug-induced gingival enlargement
4. History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
5. Anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam
6. Systemic antibiotic therapy during the 3 months preceding the baseline exam,
7. Taking immunosuppressant medications
8. Known allergy to local anaesthetic
9. History of alcohol or drug abuse
10. Self-reported pregnancy or lactation
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that according to the investigator may increase the risk associated with trial participation
12. Periodontal treatment to the study site within the last 12 months (excluding not-extensive subgingival debridement as judged by the examining clinician).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic whole defect depth reduction | 12 months
  Radiographic whole defect depth reduction in millimeters at 12 months [considered a surrogate measure evaluating the entire regenerative process including bone, cementum and periodontal ligament (Polimeni et al. 2009)]

SECONDARY OUTCOMES:
Probing Pocket Depth change | 12 months
  Probing Pocket Depth (PPD) change (in mm) at 12 months
Clinical Attachment Level change | 12 months
  Clinical Attachment Level (CAL) change at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, DipDent, MSc, PhD, Principal Investigator — Barts & The London School of Medicine & Dentistry, QMUL
Locations (9):
- Dr Ryan Lee Private Practice, Brisbane, Australia
- Studio Dentistico Associato Montevecchi D'Alessandro, Forlimpopoli, Italy
- Clinica de Periodoncia, A Coruña, Spain
- United Kingdom (6):
  - South Coast Dental Specialists, Dorchester
  - The Dentist, London
  - High Barnet Dental Care, London
  - Pall Mall Dental, London
  - Ravenscourt Dental Practice, London
  - Claremont Dental Practice, Middlesex

REFERENCES:
- [Background] Papapanou PN, Tonetti MS. Diagnosis and epidemiology of periodontal osseous lesions. Periodontol 2000. 2000 Feb;22:8-21. doi: 10.1034/j.1600-0757.2000.2220102.x. No abstract available. PMID 11276518
- [Background] Papapanou PN, Wennstrom JL. The angular bony defect as indicator of further alveolar bone loss. J Clin Periodontol. 1991 May;18(5):317-22. doi: 10.1111/j.1600-051x.1991.tb00435.x. PMID 2066446
- [Background] Heitz-Mayfield LJ, Trombelli L, Heitz F, Needleman I, Moles D. A systematic review of the effect of surgical debridement vs non-surgical debridement for the treatment of chronic periodontitis. J Clin Periodontol. 2002;29 Suppl 3:92-102; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.5.x. PMID 12787211
- [Background] Nyman S, Lindhe J, Karring T, Rylander H. New attachment following surgical treatment of human periodontal disease. J Clin Periodontol. 1982 Jul;9(4):290-6. doi: 10.1111/j.1600-051x.1982.tb02095.x. PMID 6964676
- [Background] Cortellini P, Tonetti MS. Focus on intrabony defects: guided tissue regeneration. Periodontol 2000. 2000 Feb;22:104-32. doi: 10.1034/j.1600-0757.2000.2220108.x. No abstract available. PMID 11276509
- [Background] Needleman IG, Worthington HV, Giedrys-Leeper E, Tucker RJ. Guided tissue regeneration for periodontal infra-bony defects. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD001724. doi: 10.1002/14651858.CD001724.pub2. PMID 16625546
- [Background] Trombelli L, Farina R, Franceschetti G, Calura G. Single-flap approach with buccal access in periodontal reconstructive procedures. J Periodontol. 2009 Feb;80(2):353-60. doi: 10.1902/jop.2009.080420. PMID 19186978
- [Background] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402
- [Background] Nibali L, Pometti D, Tu YK, Donos N. Clinical and radiographic outcomes following non-surgical therapy of periodontal infrabony defects: a retrospective study. J Clin Periodontol. 2011 Jan;38(1):50-7. doi: 10.1111/j.1600-051X.2010.01648.x. Epub 2010 Nov 22. PMID 21091528
- [Background] Ribeiro FV, Casarin RC, Palma MA, Junior FH, Sallum EA, Casati MZ. Clinical and patient-centered outcomes after minimally invasive non-surgical or surgical approaches for the treatment of intrabony defects: a randomized clinical trial. J Periodontol. 2011 Sep;82(9):1256-66. doi: 10.1902/jop.2011.100680. Epub 2011 Feb 2. PMID 21284549
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238
- [Derived] Mehta J, Montevecchi M, Garcia-Sanchez R, Onabolu O, Linares A, Eriksson F, Ghezzi C, Donghi C, Lu EM, Nibali L. Minimally invasive non-surgical periodontal therapy of intrabony defects: A prospective multi-centre cohort study. J Clin Periodontol. 2024 Jul;51(7):905-914. doi: 10.1111/jcpe.13984. Epub 2024 May 6. PMID 38710583